CLINICAL TRIAL: NCT01507168
Title: A Randomised, Placebo-controlled, Double-blind, Multicenter Phase II Trial of Intravenous GC33 at 1600 mg Q2W in Previously Treated Patients With Unresectable Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: A Study of GC33 (RO5137382) in Patients With Advanced or Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP27884; 2011-003574-84 (EudraCT Number)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — codrituzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GC33 (RO5137382) (Experimental)
  Interventions: Drug: GC33

INTERVENTIONS:
Drug: Placebo — iv Days 1 and 8, and every 2 weeks thereafter
  Arms: Placebo
Drug: GC33 — 1600 mg iv Day 1 and 8, and every 2 weeks thereafter
  Other Names: RO5137382
  Arms: GC33 (RO5137382)

SUMMARY:
This randomized, placebo-controlled, multicenter study will evaluate the efficacy and safety of GC33 (RO5137382) in previously treated patients with unresectable advanced or metastatic hepatocellular carcinoma. Participants will be stratified according to the level of GPC-3 expression in tumors and randomized to receive either GC33 (1600 mg intravenously) or placebo on Days 1 and 8 of Cycle 1 and every 2 weeks thereafter. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed hepatocellular carcinoma (without fibro-lamellar subtype)
* Prior treatment with at least 1 systemic agent, with documented progressive disease after systemic agent(s), or documented adverse event(s) associated with prior systemic agent(s) that resulted in discontinuance of that (those) agent(s)
* Not a candidate for curative treatments (e.g. resection, transplantation)
* Child-Pugh A (score of 5-6)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic, hepatic and renal function
* Ability to provide, for central review, a tumor tissue sample to determine the level of GPC-3 expression by IHC
* Measurable disease by RECIST criteria

Exclusion Criteria:

* Child Pugh B or C
* Known hepatocellular carcinoma with fibro-lamellar histology
* Known brain or leptomeningeal metastases
* Active infectious diseases requiring treatment except for hepatitis B and C
* History of organ allograft including liver transplant
* Anticipated or ongoing administration of anticancer therapies other than those administered in this study
* Anticancer treatment within 2 weeks prior to entering the study
* Patients who have not fully recovered from toxicities associated with previous HCC loco-regional or systemic therapies
* Patients receiving interferon therapy
* Pregnant or lactating women
* Known HIV positivity or AIDS-related illness
* History of significant hypersensitivity to similar agents (monoclonal antibody, protein-included drugs, Chinese hamster ovary products)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (tumor assessments according to RECIST criteria) | approximately 24 months

SECONDARY OUTCOMES:
Overall survival | approximately 32 months
Time to progression (TTP): Time from randomization to first documented disease progression | approximately 24 months
Disease control rate (DCR): Complete response, partial response or stable disease lasting at least 6 weeks | approximately 24 months
Safety: Incidence of adverse events | approximately 24 months
Pharmacokinetics: Serum concentrations (Cmax,Cmin) | Multiple sampling pre- and post-dose Days 1 and 8 Cycle 1, Day 1 Cycle 6, pre-dose Day 1 Cycles 2-11
GPC-3 expression in tumor tissue (biopsy) by immunohistochemistry (IHC) assay | at screening

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- United States (8):
  - UCLA Medical Center, Los Angeles, California
  - National Cancer Institute; Ctr for Cancer Research, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington Univ School of Med; Barnes-Jewish Hospital; Siteman Cancer Center, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Swedish Cancer Inst., Seattle, Washington
- Belgium (2):
  - Hospital Erasme, Brussels
  - UZ Gent, Ghent
- France (7):
  - Hotel Dieu; Medecine A, Angers
  - CHU de GRENOBLE; UF de Cancérologie, Grenoble
  - Aphm; Hopital De La Conception, Marseille
  - Hopital de L'Archet; Pole de Reference Hepatite C, Nice
  - Hôpital Saint Antoine; Service Hépathologie, Paris
  - Hopital Purpan;Gastro Enterologie Hepatologie, Toulouse
  - Hôpital d'Adultes; Service hépato-gastro-entérologie, Vandœuvre-lès-Nancy
- Germany (5):
  - Charité Uni.-medizin Berlin, Campus Virchow-Klinikum; Med. Klinik m.S. Hepatologie Gastroenterologie, Berlin
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik I, Frankfurt am Main
  - Uni Heidelberg Med. Klinik; Innere Medizin IV, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der TU München; Klinikapotheke, München
- Hong Kong (2):
  - Queen Mary Hospital; Dept of Surgery, Pokfulam
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (3):
  - Azienda Ospedaliera G. Rummo; Unità Operativa di Oncologia Medica 1, Benevento, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione IRCCS Ospedale Maggiore Policlinico; Gastroenterologia, Milan, Lombardy
- Japan (6):
  - National Cancer Center Hospital East, Chiba
  - Kanazawa University Hospital, Ishikawa
  - Kanagawa Cancer Center, Kanagawa
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
- Auckland Hospital; New Zealand Liver Transplant Unit, Auckland, New Zealand
- National Cancer Centre; Medical Oncology, Singapore, Singapore
- South Korea (6):
  - Pusan University Hospital, Busan
  - National Cancer Center, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (8):
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron; Servicio de Hepatologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario Miguel Servet; Servicio Hematologia, Zaragoza
- Taiwan (5):
  - Chang Gung Memorial Foundation - Kaohsiung, Kaohsiung City
  - Taichung Veterans Gen Hosp, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - The Clatterbridge Cancer Ctr NHS Foundation Trust, Bebington
  - Royal Free Hospital; Dept of Oncology, London
  - King'S College Hospital; Haematology, London

REFERENCES:
- [Derived] Pradier MF, Reis B, Jukofsky L, Milletti F, Ohtomo T, Perez-Cruz F, Puig O. Case-control Indian buffet process identifies biomarkers of response to Codrituzumab. BMC Cancer. 2019 Mar 28;19(1):278. doi: 10.1186/s12885-019-5472-0. PMID 30922327
- [Derived] Abou-Alfa GK, Puig O, Daniele B, Kudo M, Merle P, Park JW, Ross P, Peron JM, Ebert O, Chan S, Poon TP, Colombo M, Okusaka T, Ryoo BY, Minguez B, Tanaka T, Ohtomo T, Ukrainskyj S, Boisserie F, Rutman O, Chen YC, Xu C, Shochat E, Jukofsky L, Reis B, Chen G, Di Laurenzio L, Lee R, Yen CJ. Randomized phase II placebo controlled study of codrituzumab in previously treated patients with advanced hepatocellular carcinoma. J Hepatol. 2016 Aug;65(2):289-95. doi: 10.1016/j.jhep.2016.04.004. Epub 2016 Apr 13. PMID 27085251